CLINICAL TRIAL: NCT05403034
Title: Study of the Biological Function of Muscle Satellite Cells From Patients With Obstetric Brachial Plexus Palsy Satellite Cell Obstetrical PlExus (SCOPE)
Brief Title: Study of the Biological Function of Muscle Satellite Cells From Patients With Obstetric Brachial Plexus Palsy
Acronym: SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL21_0524; 2021-A02669-32 (Other: number IDRCB)
Record Dates: First submitted 2022-04-26; First posted 2022-06-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Obstetrical Brachial Plexus Palsy
Keywords: Brachial plexus; Neonatal brachial plexus palsy; Denervation; Muscle atrophy; Muscle regeneration; Botulinum toxin; Satellite cell; Primary human muscle cell culture
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OBPP children (Experimental): OBPP children operated on to treat shoulder stiffness.
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — Peroperative muscle biopsy will be performed during a planned shoulder surgery (arthrolysis and/or muscle transfer)
  Other Names: Shoulder arthrolysis; Shoulder muscle transfer

SUMMARY:
The purpose of this prospective work is to study the consequences of obstetrical brachial plexus paralysis on the rotator muscles of the shoulder. The hypothesis is that shoulder stiffness of these children is due to an impairment of the shoulder rotator muscles. The investigators want to test the regenerative capacities of these muscles. The development of a cellular model of this pathology will allow to test new therapeutic perspectives and to validate our hypothesis.

DETAILED DESCRIPTION:
During delivery, there can be a lesion of the nerve roots of the brachial plexus (cervical C5-C8 and/or thoracic T1 roots). The newborn presents at birth a paralysis of the arm (Obstetrical Brachial Plexus Paralysis: OBPP). One third of children with OBPP will have sequelae despite daily rehabilitation. The most frequent disability is shoulder stiffness. The current hypothesis is that this stiffness is due to a permanent imbalance between the affected shoulder muscles (lateral rotators) and the muscles less affected by the paralysis (medial rotators). Because of this imbalance, the injured shoulder is spontaneously positioned in medial rotation. This position would lead to retractions at the front of the joint despite rehabilitation. In case of incomplete recovery, growth disorders of the shoulder joint (dysplasia) appear as well as a functional handicap.

The management, from the age of 2 years, in case of shoulder stiffness and dysplasia, is surgery (arthrolysis) to regain mobility. During this operation, a muscle transfer can also be performed to strengthen the lateral rotator muscles.

However, despite surgery, mobility deficits often recur within a few years. To understand the origin of the lateral and medial rotation deficits, the investigators conducted an anatomopathological study of the rotator muscles in these children. The preliminary results show a significant damage of the rotator muscles with the presence of fibrosis which could explain the rotational stiffness and the functional impairment. To better understand the pathophysiological mechanisms, the investigatorswill set up an OBPP model in cell culture to understand the regenerative capacities and to test new pharmacological approaches.

ELIGIBILITY:
Inclusion Criteria:

* OBPP children with a planned shoulder surgery (arthrolysis and/or muscle transfer).

Exclusion Criteria:

* other neurological disorders, post-traumatic shoulder stiffness

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Assessment of muscle regeneration capacity: proliferation capacity | 30 days
  Proliferation capacity of satellite cells assessed by immunofluorescence: percentage of Pax 7 positive cells/total desmin positive cells
assessment of muscle regeneration capacity: differenciation capacity | 30 days
  Differentiation capacity of satellite cells assessed by histology: fusion index (number of nuclei in a myotubule compared to total number of nuclei in the sample) in percentage

SECONDARY OUTCOMES:
Effect of botulinum toxin on the proliferation potential of satellite cells: proliferation capacity | 30 days
  Proliferation capacity of satellite cells assessed by immunofluorescence: percentage of Pax 7 positive cells/total desmin positive cells.
Effect of botulinum toxin on the proliferation potential of satellite cells: differentiation capacity | 30 days
  Differentiation capacity of satellite cells assessed by histology: fusion index (number of nuclei in a myotubule compared to total number of nuclei in the sample) in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Marion DELPONT, Dr, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Chu Montpellier, Montpellier, France